CLINICAL TRIAL: NCT03622099
Title: Transthoracic Echocardiography Guided Small Volume Fluid Challenge as a Predictor of Fluid Responsiveness in Patients With Circulatory Failure: An Observational Study
Brief Title: Small Volume Fluid Challenge as a Predictor of Fluid Responsiveness in Patients With Circulatory Failure
Status: Completed | Type: Observational
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Abd-Elazeem Abd-Elhameed Elbakry, Assistant professor, Menoufia University
Other Study IDs: 2017/3/1/4
Record Dates: First submitted 2018-07-30; First posted 2018-08-09 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Circulatory Failure
MeSH Terms: conditions — Shock | interventions — Saline Solution

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study group: As a routine work in adult critical care unit at Menoufia University hospital for patients with circulatory failure, A 100 ml bolus of Normal Saline Flush, 0.9% Injectable Solution was given to the patient over 1 minute through a central venous catheter or jugular cannula. For prediction of responders, echocardiographic parameters measured followed by infusion of the remaining 400 ml of Normal Saline Flush, 0.9% Injectable Solution at a constant rate over 10 minutes then echocardiographic parameters measured again to detect the patient response.
  Interventions: Drug: Normal Saline Flush, 0.9% Injectable Solution

INTERVENTIONS:
Drug: Normal Saline Flush, 0.9% Injectable Solution — As a routine work in adult critical care unit at Menoufia University hospital for patients with circulatory failure, A 100 ml bolus of Normal Saline Flush, 0.9% Injectable Solution was given to the patient over 1 minute through a central venous catheter or jugular cannula. For prediction of responders, echocardiographic parameters measured followed by infusion of the remaining 400 ml of Normal Saline Flush, 0.9% Injectable Solution at a constant rate over 10 minutes then echocardiographic parameters measured again to detect the patient response.
  Other Names: normal saline

SUMMARY:
Assessment of intravascular volume status is difficult in critically ill patients. Evidence suggests that only 50% of hemodynamically unstable patients respond to a fluid challenge. Moreover, if cardiopulmonary function cannot compensate for the increase in preload, fluid loading may compromise microvascular perfusion and oxygen delivery and cause or aggravate peripheral and pulmonary edema. Inappropriate fluid expansion can increase morbidity and mortality thus making it important to accurately assess fluid responsiveness in critically ill patients. The volume responsiveness can be defined as a 15% increase in stroke volume (SV) or cardiac output (CO) after a 500-ml infusion. This study tested whether echocardiographic parameters can predict fluid responsiveness in critically ill patients following a low volume 100-ml crystalloid solution infusion over 1 minute.

DETAILED DESCRIPTION:
Fifty-four adult patients with circulatory failure were recruited for the study. As a routine work in adult critical care unit at Menoufia University hospital for patients with circulatory failure, a 100 ml bolus of normal saline solution was given to the patient over 1 minute through a central venous catheter or jugular cannula. For prediction of responders, echocardiographic parameters were recorded1 minute after bolus administration. The remaining 400 ml of normal saline solution was infused at a constant rate over 10 minutes, and echocardiographic parameters were recorded again. The mean echocardiographic measurements over three consecutive respiratory cycles were recorded along with heart rate HR, systolic, diastolic and mean arterial pressures, central venous pressure, and Temperature also mechanical ventilation parameter (tidal volume, respiratory rate and PEEP) for each patient. Patients with an increase in CO after a 100 ml or total 500-ml infusion over 10 minutes (ΔCO500) of 15% or more were classified as responders (Rs) and those without an increase in CO was classified as non-responders

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute circulatory failure
* Mechanically ventilated & sedated.(Tidal volume 6-8 ml/ kg, PEEP 5 mmHg, Richmond Agitation-Sedation Scale RASS (R) Score from zero to -3).
* Systemic inflammatory response syndrome
* Septic shock
* Controlled massive hemorrhage

Exclusion Criteria:

* Age of less than 18 years
* Cardiomyopathy
* Pulmonary edema
* Morbid obesity
* Pregnancy
* Increased intracranial tension
* Valvular heart disease
* Myocardial ischemia or infarction before the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: in a general adult critical care unit (CCU) at Menoufia University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Aortic blood flow velocity Time Integral changes from the baseline | Baseline 10 minutes before start of fluid challenge and1 minute after fluid challenge
  [cm]

SECONDARY OUTCOMES:
stroke volume change from the baseline | Baseline 10 minutes before start of fluid challenge and1 minute after fluid challenge
  [ml/beat]
cardiac output change from the baseline | Baseline 10 minutes before start of fluid challenge and1 minute after fluid challenge
  [ liter/minute]
heart rate change from the baseline | Baseline 10 minutes before start of fluid challenge and1 minute after fluid challenge
  [beats/minute]
systolic blood pressure change from the baseline | Baseline 10 minutes before start of fluid challenge and1 minute after fluid challenge
  [mmHg]
Diastolic blood pressure change from the baseline | Baseline 10 minutes before start of fluid challenge and1 minute after fluid challenge
  [mmHg]
Central venous pressure change from the baseline | Baseline 10 minutes before start of fluid challenge and1 minute after fluid challenge
  [Cm water]
Mean arterial blood pressure change from the baseline | Baseline 10 minutes before start of fluid challenge and1 minute after fluid challenge
  [mmHg]
Left ventricular end systolic diameter change from the baseline | Baseline 10 minutes before start of fluid challenge and1 minute after fluid challenge
  [Cm]
Left ventricular end diastolic diameter change from the baseline | Baseline 10 minutes before start of fluid challenge and1 minute after fluid challenge
  [Cm]
Aortic root diameter change from the baseline | Baseline 10 minutes before start of fluid challenge and1 minute after fluid challenge
  [Cm]

CONTACTS AND LOCATIONS:
Overall Officials: Abd-Elazeem A Elbakry, M.D, Study Chair — Menoufia University
Locations (1):
- Faculty of Medicine, Cairo, Shebin El-kom, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the paper protocol only we share if the paper is published in a closed access journal. For open access no problem for sharing the whole data
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication
Access Criteria: through the clinical trial registry site or contact by my e-mail